CLINICAL TRIAL: NCT00004438
Title: Study of Leuprolide in Adults With Hypogonadotropism
Brief Title: Leuprolide in Treating Adults With Hypogonadotropism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13402; UCCH-8451; UCCH-FDR001473
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1998-06

CONDITIONS: Hypogonadism
Keywords: endocrine disorders; hypogonadism; rare disease
MeSH Terms: conditions — Hypogonadism; Endocrine System Diseases; Rare Diseases | interventions — Leuprolide

INTERVENTIONS:
Drug: leuprolide

SUMMARY:
RATIONALE: Hypogonadotropism is an abnormal condition caused by decreased production of gonadotropins, a group of hormones that stimulate the parts of the reproductive system that produce and release eggs from the ovaries or sperm from the testicles. Leuprolide may stimulate the production of gonadotropins and be effective in increasing testosterone in men and inducing ovulation in women.

PURPOSE: Clinical trial to study the effectiveness of leuprolide in treating adults who have hypogonadotropism.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Male patients receive leuprolide subcutaneously every 5 days for up to one year and are followed at weeks 4, 6, 8, and 12, then every 2 months.

Female patients receive leuprolide subcutaneously on days 1, 6, and possibly 11. Patients are followed 2 months after the last injection.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of hypogonadotropism

Men: Small testes, abnormal semen analysis, and subnormal plasma testosterone levels without an elevation in gonadotropin levels

Women: Amenorrhea and subnormal plasma estradiol levels, or lack of cornification of the vaginal mucosa without an elevation in gonadotropin levels OR Hypothalamic amenorrhea in normally estrogenized women with amenorrhea or oligomenorrhea and normal plasma free testosterone and gonadotropin levels

Patients with hyperprolactinemia eligible only if hypogonadotropism persists after correction of hyperprolactinemia by dopamine agonist therapy

--Prior/Concurrent Therapy-- At least 2 months since sex hormone treatment

--Patient Characteristics--

Other:

* Not pregnant
* No chronic systemic, metabolic, or endocrine disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 1997-09; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Rosenfield, Study Chair — University of Chicago
Locations (1):
- University of Chicago Children's Hospital, Chicago, Illinois, United States